CLINICAL TRIAL: NCT02577965
Title: Optical Coherence Tomography Assessment of Gender diVersity In Primary Angioplasty: The OCTAVIA Trial
Acronym: OCTAVIA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A.O. Ospedale Papa Giovanni XXIII (Other)
Collaborators: Light Lab Imaging, Inc. (Industry)
Responsible Party: Principal Investigator, GGuagliumi, MD, A.O. Ospedale Papa Giovanni XXIII
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5/01/2011-2
Record Dates: First submitted 2014-09-15; First posted 2015-10-16 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Acute Myocardial Infarction
Keywords: ST segment Elevation Myocardial Infarction; Optical Coherence Tomography; Percutaneous Coronary Intervention; Thrombus histopathology; Gender differences
MeSH Terms: conditions — ST Elevation Myocardial Infarction | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Female Arm (Experimental): Female gender diagnosed with ST segment Elevation Myocardial Infarction (STEMI). Interventions: Angiography, thrombus aspiration, optical coherence tomography and percutaneous coronary intervention, implantation of XIENCE PRIME Everolimus Eluting Coronary Stent. Angiography and Optical Coherence Tomography follow up at 9 months.
  Interventions: Procedure: Percutaneous Coronary Intervention; Device: XIENCE PRIME Everolimus Eluting Coronary Stent System
- Male Arm (Active Comparator): Male Gender with diagnose of ST segment Elevation Acute Myocardial Infarction (STEMI). Interventions: Angiography, thrombus aspiration, optical coherence tomography and percutaneous coronary intervention, implantation of XIENCE PRIME Everolimus Eluting Coronary Stent. Angiography and Optical Coherence Tomography follow up at 9 months.
  Interventions: Procedure: Percutaneous Coronary Intervention; Device: XIENCE PRIME Everolimus Eluting Coronary Stent System

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention — Thrombus aspiration and histopathological analysis ,Optical Coherence Tomography assessment of culprit vessel during primary PCI, Primary PCI and Drug Eluting Stent (DES) - XIENCE PRIME Everolimus Eluting Coronary Stent implantation in culprit lesion, coronary angiography and OCT assessment at 9 months follow-up
Device: XIENCE PRIME Everolimus Eluting Coronary Stent System — Xience Prime Everolimus Eluting Coronary Stent System implantation to treat Acute Myocardial Infarction

SUMMARY:
Recent studies suggest important gender differences in the pathophysiology and prognosis of ST-segment elevation myocardial infarction (STEMI). This is the first prospective controlled study to assess gender differences in the mechanism of plaque rupture/erosion and thrombus formation in patients presenting with STEMI treated with primary angioplasty. Gender-related mechanisms of plaque rupture or erosion will be investigated using a combination of Quantitative Coronary Angiography (QCA), high resolution Optical Coherence Tomography (OCT) of the culprit vessel and histopathology analyses of thrombus aspirates of the infarct related lesion, performed by independent core laboratories, blinded to group (male or female) and clinical variables.

In OCTAVIA; enrollment in a 1:1 ratio according to gender group will be ensured by a computer-assisted matching algorithm for gender and age (< 50, 51-70, and > 70 years). Matching has the purpose to enable enrollment of an even number of male and female patients in balanced age groups. This type of dynamic algorithm is appropriate when the composition of the referral population is not known in advance.

The sample size for the OCTAVIA study was calculated on the basis of per patient stent strut coverage (a continuous variable with right skewed distribution) with mean of 97.0% and standard deviation of 4.0% in men, versus mean of 95.0% and standard deviation of 4.0% in women, following XIENCE PRIME™ Everolimus Eluting Coronary Stent System implantation. Thus, aiming for a 5% 2-tailed superiority alpha, an 80% power, and assuming a 1:1 enrollment according to gender, a total of 64 patients per group should be enrolled. Anticipating a 10% dropout rate due to patients lost to follow-up and inadequate imaging (included major side branch sections), the total enrollment is set at 70 patients per group (total population of 140 subjects).

DETAILED DESCRIPTION:
A suboptimal degree of attention has focused on the detection and management of coronary artery disease (CAD) in women until recently. Although many women do not perceive heart disease as a significant health risk, CAD is the leading cause of mortality in women in most developed nations, with mortality primarily driven by acute ST-elevation myocardial infarction (STEMI) and cardiogenic shock (American Heart Association 2005 Heart Disease and Stroke Statistics).

In recent years, literature articles regarding various aspects of heart disease in women significantly increased. These reports have highlighted important sex differences in the pathophysiology, presentation, and treatment of ischemic heart disease and have denounced pervasive sex-related disparities in referral and treatment for heart disease as a major reason for outcome differences between the sexes. Such activities have been useful in driving attention to heart disease in women, an area largely ignored by the scientific community and the public just 20 years ago.

However, we must recognize that to date, limited data substantiate many of these statements; such recognition is important to guide future research efforts. A careful look at recently published literature reveals only modest advancements toward clarifying gender-based differences in the pathophysiology of ischemic heart disease and gender-based differences in outcome. At the same time, key questions concerning strategies for prevention and treatment of heart disease in women remain unanswered, and cardiovascular clinical trials continue to include fewer women than men.

A fundamental question is whether the mechanisms underlying ischemic heart disease in women differ from those in men. This is an important question because if pathophysiology differs in women, such differences can inform strategies for prevention, detection, and treatment that would be most effective for women.

A number of indicators point to a different mechanism in man and women.

1. More symptoms, but less diseased vessels. Despite having more symptoms and physical limitations, women have less obstructive coronary heart disease than men, as assessed by angiography along the entire spectrum of acute coronary syndromes. Chest pain without apparently severe obstructive coronary artery disease (CAD) is distinctly more common in women than in men.
2. Disability unrelated to severity of coronary obstructions. Among women, chest pain symptoms and disability do not correlate with severity of coronary stenosis, assessed by angiography.
3. Higher risk after infarction despite lesser cardiac damage. Women, particularly those who are young or middle-aged (whom one would expect to be most advantaged for coronary disease risk compared with men due to estrogen protective actions), show higher rates of adverse outcomes after acute myocardial infarction (MI) than men of similar age, despite less severe coronary narrowing, smaller infarcts, and more preserved systolic function.

Consequently, the identification of less obstructive atheroma has been put forth as a potentially helpful strategy for the risk stratification of women.

Although this is a compelling theory, to date there is little evidence to suggest that vascular abnormalities in the absence of obstructive atheroma as detected by angiography are more commonly implicated in the pathogenesis of ischemia among women than men.

Recent studies have evaluated gender differences in coronary structure and function using intravascular ultrasound and other types of vascular testing. These studies have found that women had less atheroma volume than men, including both luminal plaque and atheroma within the media, despite older age and more risk factors, and even after accounting for body surface area and vessel size. After adjusting for body size, women also have smaller coronary vessels. However, these studies were unable to identify other vascular abnormalities, like plaque characteristics, that might explain gender differences in clinical presentation.

Presently, we are far from being able to conclude, or even suggest, that these hypothesized abnormalities play a larger etiologic or prognostic role for ischemic heart disease among women than among men.

A general pattern of higher mortality and complication rates in women after acute coronary syndromes (ACS) compared with men has been described for many years. It is important to recognize, however, that gender differences in mortality after ACS do not occur across the board but only in specific patient subgroups.

It is hypothesized that differences by MI type (STEMI versus other types) may be due to the pathophysiology underlying these events. For example, acute occlusion caused by thrombus superimposed on a ruptured or eroded atherosclerotic plaque is believed to play a larger role in trans mural infarctions than other types of ACS. Thus, it is possible that gender differences in vessel size and collateralization put women at greater risk than men after STEMI but not after other types of ACS.

It is also unclear why gender differences in the outcome of MI are seen in young and middle-aged patients but not older patients. One would expect that women younger than 50 years of age, the majority of whom are premenopausal, should be more advantaged rather than less advantaged compared with men of similar age in terms of survival. On the other hand, for coronary disease to occur in younger women, it must be aggressive, driven by multiple risk factors, or caused by secondary or unknown causes.

A less aggressive clinical treatment of women with coronary heart disease relative to men has been documented for years, with a tendency to refer to it as gender bias in health care delivery.

A 2005 Statement from the American Heart Association reviewed gender-specific data on the safety and efficacy of percutaneous coronary intervention and pharmacotherapy. Despite the fact that more women than men die from cardiovascular disease in the United States, and despite the established benefits of Percutaneous Coronary Intervention (PCI) in reducing fatal and nonfatal ischemic complications in patients with acute myocardial infarction, only an estimated 33% of annual PCIs are performed in women. In addition, women experience greater delays to intervention and are referred for diagnostic catheterization less frequently than are men.

Recent advances in angioplasty equipment and technique have improved options for patients with smaller coronary and peripheral (access) arteries. In addition, the increased use of stents and adjunctive pharmacotherapy has improved outcomes in both women and men. Nevertheless, women continue to represent 15% to 38% of the population in studies of PCI, and still relatively few gender- or race-specific data exist.

According to the American Heart Association, better understanding and elimination of this apparent treatment disparity is a priority. One of the areas of interest is to refine treatment pathways and strategies for women with STEMI, in whom mortality rates and bleeding risk remain higher than in men.

To further optimize clinical outcomes of women undergoing PCI, evidence-based evaluation in randomized clinical trials must emphasize increased recruitment of women, with mandates to include gender-specific, ethnic, and racial gender-based results.

Cardiovascular Optical Coherence Tomography (OCT) is an innovative catheter-based imaging technology that utilizes light rather than ultrasound to obtain unique details of the vessels on a microscopic scale. OCT provides high-resolution (10 to 15 micron axial), full tomographic in vivo images and measurements of coronary arteries and deployed stents with a high level of accuracy.(8,9) Applications of this technique include diagnostic assessments of coronary atherosclerosis and guidance of coronary interventions.

After at least a decade of renewed interest in women's cardiovascular health, we are left with more questions than answers. Fundamental questions about the pathophysiology of ischemic heart disease in women remain unanswered. We have gained few clues about the basis for gender differences in coronary heart disease and what is unique about the female vascular system. As a result, we are yet unable to explain gender differences in the epidemiology, presentation, treatment and outcome of coronary heart disease. Key questions remain about why women are protected from cardiovascular disease, why this protection is restricted to the coronary system, and why this protection ends when women have diabetes or an acute MI.

We lack studies that compare biological mechanisms of disease between women and men to better define vascular processes that are unique to women. We lack sufficiently large follow-up studies to link such processes to cardiac end points. How can we increase the inclusion of women in cardiovascular clinical trials? Without an answer to these questions, little can be done to improve the prevention and the treatment of coronary heart disease in women.

In STEMI patients, acute coronary occlusion caused by thrombus superimposed on a ruptured or eroded plaque plays an important role. Nevertheless, no evidence is available concerning the mechanism of plaque rupture, the underlying vascular abnormalities of the infarct related vessel and the biological responses such as vascular remodeling and repair, that are unique to women.

In the OCTAVIA trial, gender-related mechanisms of plaque rupture will be investigated using a combination of Quantitative Coronary Angiography (QCA), OCT and histopathology analyses of thrombus aspirates of the culprit lesion performed by independent core laboratories, blinded to the group assignment.

By combining clinical variables with QCA, OCT and thrombus analysis, it is possible to obtain critical information concerning the relationship between serological biomarker of cardiac damage, clinical and prognostic correlates of coronary plaque morphology and the underlying mechanisms of coronary thrombosis in women.

In addition to assessing gender differences in the mechanism of plaque rupture, OCTAVIA will also evaluate the changes in the vascular territory remote from the infarct related lesion, the local vascular response to primary angioplasty interventions and the correlation with clinical outcomes over one year of follow-up. These data are important to support a gender based differential strategy and can have a substantial impact for the improvement of clinical practice in the treatment of women with STEMI.

ELIGIBILITY:
Inclusion Criteria:

* Acute Myocardial MI with ST segment Elevation, within 6 hours from symptoms onset
* Native coronary artery disease (no prior stent implant, no prior brachytherapy)
* Signed patient informed consent

Exclusion Criteria:

* Patients with left main disease
* infarct lesions in bypass grafts
* cardiogenic shock
* renal failure
* recent major bleeding
* allergy to aspirin or clopidogrel
* on anticoagulant therapy
* no suitable anatomy for OCT (extreme tortuousity, very distal culprit lesion, and large infarct vessel > 4 mm in diameter)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
percentage of ruptured or eroded plaques at infarct related lesion as assessed by OCT before PCI | within 6 hours from symptoms onset
  To assess gender differences in the percentage of ruptured or eroded plaques at infarct related lesion as assessed by OCT before PCI.

SECONDARY OUTCOMES:
Minimal Fibrous Cap Thickness (µm) at infarct-related lesion. | within 6 hours from symptoms onset
  To assess gender differences in Minimal Fibrous Cap Thickness at infarct related lesion.
Presence and type of thrombus at culprit site | within 6 hours from symptoms onset
  To assess gender differences in thrombus type at culprit site
Number of Thin Cat Fibroatheroma (TCFA) (<65 µM) in the scanned segment. | within 6 hours from symptoms onset
  To assess gender difference in TCFA number in culprit site
percent of incompletely apposed-uncovered struts | 9 months
  to assess gender difference in % incompletely apposed/uncovered struts at 9 months follow up by OCT
percent net volume obstruction | 9 months
  To assess gender difference in % of stent volume obstruction by OCT at 9 months follow up
percent abnormal intraluminal tissue | 9 months
  To assess gender difference in % of abnormal intraluminal tissue by OCT at 9 months follow up
percent of covered stent struts by OCT | 9 months
  To assess gender differences in the percentage of covered stent struts by OCT at 9 months follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Giulio Guagliumi, MD, Principal Investigator — Italian Society of Interventional Cardiology (GISE)